CLINICAL TRIAL: NCT05112614
Title: Role of Gut Microbiome in Cancer Therapy
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 19-003060; NCI-2021-10793 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-10-22; First posted 2021-11-09 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (biospecimen collection, medical record review): Patients undergo collection of blood and stool samples and have their medical records reviewed.
  Interventions: Procedure: Biospecimen Collection; Other: Electronic Health Record Review

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood and stool samples
  Other Names: Biological Sample Collection; Biospecimen Collected
Other: Electronic Health Record Review — Review of medical records

SUMMARY:
This study examines how gut microbiome can affect cancer therapy in cancer patients undergoing cancer therapy or stem cell transplant. The human microbiome affects the way some cancer drugs are metabolized in the human body. Information from this study may help doctors improve the way cancer treatment is delivered, and increase its effectiveness and success.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To correlate gut microbiome with specific cancer diagnoses and the clinical response (efficacy), and adverse effects of cancer therapy (single or multiple) and stem cell transplant.

OUTLINE:

Patients undergo collection of blood and stool samples and have their medical records reviewed.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-99
* Diagnosis of cancer and undergoing cancer therapy or scheduled to start cancer therapy or undergoing stem cell transplant for any hematological condition

Exclusion Criteria:

* Unable to provide informed consent
* Vulnerable adults

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cancer therapy for any underlying cancer diagnosis and patients undergoing stem cell transplant for any hematological condition
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2019-09-11 (Actual); Primary Completion 2029-10-01 (Estimated); Study Completion 2030-10-01 (Estimated)

PRIMARY OUTCOMES:
Gut microbiome associations with cancer diagnoses | Through study completion, average of 1 year
  Will be done using Shogun pipeline for metagenomics data followed by analysis using QIIME 2.0.
Associations between microbial community abundances and clinical outcomes | Through study completion, average of 1 year
  Will use a linear multivariate regression model specifically developed for microbiome data (MaAsLin, Multivariate microbial Association by Linear models.

CONTACTS AND LOCATIONS:
Overall Officials: Purna C. Kashyap, MBBS, Principal Investigator — Mayo Clinic in Rochester
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials